CLINICAL TRIAL: NCT02889393
Title: Teduglutide for Treatment of Enterocutaneous Fistula (ECF) - a Pilot Study to Demonstrate Safety and Feasibility
Brief Title: Teduglutide for Enterocutaneous Fistula (ECF)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Daniel Dante Yeh (Other)
Collaborators: Takeda (Industry)
Responsible Party: Sponsor-Investigator, Daniel Dante Yeh, Associate Professor of Surgery, University of Miami
Organization: University of Miami (Other)
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: 20170189
Record Dates: First submitted 2016-08-31; First posted 2016-09-05 (Estimated); Results first posted 2021-10-06 (Actual); Last update posted 2021-10-06 (Actual); Status verified 2021-09

CONDITIONS: Postoperative Fistula
MeSH Terms: interventions — teduglutide; ALX-0600; Standard of Care

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Standard of Care followed by Teduglutide (Experimental): Participants in this group will receive standard of care treatment for the first 8 weeks followed by daily Teduglutide for the next 8 weeks.
  Subjects with a favorable response will be offered an open label extension during which they will continue to receive teduglutide for up to another 12 months or permanent fistula closure.
  Interventions: Drug: Teduglutide; Other: Standard of Care
- Teduglutide followed by Standard of Care (Experimental): Participants in this group will receive daily Teduglutide treatment for the first 8 weeks followed by standard of care for the next 8 weeks.
  Subjects with a favorable response will be offered an open label extension during which they will continue to receive teduglutide for up to another 12 months or permanent fistula closure
  Interventions: Drug: Teduglutide; Other: Standard of Care

INTERVENTIONS:
Drug: Teduglutide — Daily 0.05 mg/kg Teduglutide administered subcutaneously.
  Other Names: Gattex
Other: Standard of Care — The standard of care treatment of ECF which includes meticulous wound care, optimizations of nutrition, use of acid-suppression medications and anti-motility agents as per treating physician discretion.

SUMMARY:
The purpose of this study is to determine whether Teduglutide is safe and feasible to be given for the treatment of enterocutaneous fistula (ECF). The hypothesis is that the drug will be well tolerated and will improve the volume of daily ECF output as well as improve the functional quality of life.

ELIGIBILITY:
Inclusion Criteria:

* Age >18
* Enterocutaneous fistula (ECF) that could be secondary to volvulus, injury, prior trauma or surgery, or vascular ischemia

Exclusion Criteria:

* Perianal fistula
* Clinical suspicion of inflammatory bowel disease
* History of radiation enteritis or sprue (as defined by history)
* Active (<1 year) alcohol or drug abuse
* Significant hepatic, or cardiac diseases as defined as:
* Hepatic: aspartate aminotransferase (AST) > 2 times upper limit of normal (10-40 U/L)
* Cardiac: unstable angina or evidence of active myocardial ischemia (elevated troponin level drawn by clinical suspicion)
* Severe renal dysfunction: serum creatinine > 2 times upper limit of normal (0.6-1.5 mg/dL)
* Received glutamine less than 4 weeks prior to screening
* Receiving growth factors (erythropoietin, granulocyte colony-stimulating factor, granulo-cyte-macrophage colony stimulating factor, and human growth hormone)
* Pregnancy or lactation (women of childbearing age will be excluded if they do not agree to either complete sexual abstinence during the study or if they refuse to use at least two forms of highly effective contraception such as oral contraception, injectable or implantable contraception, vaginal rings, or intrauterine devices (IUD))
* Active malignancy or suspicion for gastrointestinal malignancy on CT scan
* Not capable of understanding or not willing to adhere to the study visit schedule and drug administration requirements
* Family history of intestinal malignancy (gastric, small intestine, colon)
* Personal or family history of hereditary non-polyposis colorectal cancer, familial adenomatous polyposis, first degree relative with colon cancer
* Positive hemoccult (per rectum)
* Abnormal baseline electrocardiogram (ECF) suggestive of congestive heart failure or underlying cardiac disease
* Taking oral benzodiazepines, barbiturates, or phenothiazines

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2019-01-31 (Actual); Primary Completion 2020-07-15 (Actual); Study Completion 2021-07-15 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Daniel D Yeh, MD, Principal Investigator — University of Miami
Locations (1):
- University of Miami, Miami, Florida, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Jeppesen PB, Lund P, Gottschalck IB, Nielsen HB, Holst JJ, Mortensen J, Poulsen SS, Quistorff B, Mortensen PB. Short bowel patients treated for two years with glucagon-like Peptide 2: effects on intestinal morphology and absorption, renal function, bone and body composition, and muscle function. Gastroenterol Res Pract. 2009;2009:616054. doi: 10.1155/2009/616054. Epub 2009 Aug 20. PMID 19707516
- [Background] Jeppesen PB, Gilroy R, Pertkiewicz M, Allard JP, Messing B, O'Keefe SJ. Randomised placebo-controlled trial of teduglutide in reducing parenteral nutrition and/or intravenous fluid requirements in patients with short bowel syndrome. Gut. 2011 Jul;60(7):902-14. doi: 10.1136/gut.2010.218271. Epub 2011 Feb 11. PMID 21317170
- [Derived] Yeh DD, Vasileiou G, Abdul Jawad K, Pust GD, Byers PM. Teduglutide for the treatment of low-output enterocutaneous fistula - A pilot randomized controlled study. Clin Nutr ESPEN. 2022 Aug;50:49-55. doi: 10.1016/j.clnesp.2022.04.031. Epub 2022 May 12. PMID 35871951

RESULTS

PARTICIPANT FLOW:
Groups:
- Standard of Care Followed by Teduglutide: Participants in this group will receive standard of care treatment for the first 8 weeks followed by daily Teduglutide for the next 8 weeks.
  Subjects with a favorable response will be offered an open label extension during which they will continue to receive teduglutide for up to another 12 months or permanent fistula closure.
  Teduglutide: Daily 0.05 mg/kg Teduglutide administered subcutaneously.
  Standard of Care: The standard of care treatment of ECF which includes meticulous wound care, optimizations of nutrition, use of acid-suppression medications and anti-motility agents as per treating physician discretion.
- Teduglutide Followed by Standard of Care: Participants in this group will receive daily Teduglutide treatment for the first 8 weeks followed by standard of care for the next 8 weeks.
  Subjects with a favorable response will be offered an open label extension during which they will continue to receive teduglutide for up to another 12 months or permanent fistula closure
  Teduglutide: Daily 0.05 mg/kg Teduglutide administered subcutaneously.
  Standard of Care: The standard of care treatment of ECF which includes meticulous wound care, optimizations of nutrition, use of acid-suppression medications and anti-motility agents as per treating physician discretion.
Period: Overall Study
Arm/Group | Standard of Care Followed by Teduglutide | Teduglutide Followed by Standard of Care
Started | 3 | 3
Completed | 3 | 3
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Standard of Care Followed by Teduglutide | Teduglutide Followed by Standard of Care | Total
Number analyzed (Participants) | 3 | 3 | 6
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 3 | 2 | 5
  >=65 years | 0 | 1 | 1
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 2 | 2
  Male | 3 | 1 | 4
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 1 | 2
  Not Hispanic or Latino | 2 | 2 | 4
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 1 | 0 | 1
  White | 2 | 3 | 5
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Change in Average 3-day Fistula Percent Volume
Description: Percent fistula volume will be reported from the participant
Time Frame: Baseline, Up to 8 weeks
Population: This is a cross-over study. Each participant received both teduglutide intervention and the standard of care intervention for 8 weeks each.
Measure: Mean (Standard Deviation); unit: Percent change in fistula volume
Groups:
- Teduglutide Intervention: Participants that received Teduglutide for 8 weeks
- Standard of Care Intervention: Participants that received Standard of Care for 8 weeks
Arm/Group | Teduglutide Intervention | Standard of Care Intervention
Number analyzed (Participants) | 6 | 6
Percent change in fistula volume | 76.33 (355.36) | 441.67 (824.87)

2. Secondary Outcome: Number of Participants With Ceased Fistula Output
Description: As evaluated by treating physician of having at least 1 ceased fistula output
Time Frame: Up to 16 weeks
Population: Ceased fistula output was reported for all participants at the end of treatment after receiving both interventions.
Measure: Count of Participants; unit: Participants
Groups:
- All Participants: Participants that received both standard of care and teduglutide interventions after a combined 16 weeks
Arm/Group | All Participants
Number analyzed (Participants) | 6
Participants | 3

3. Secondary Outcome: Quality of Life as Measured by ASCQ-Me® v2.0 Social Functioning - Short Form
Description: Adult Sickle Cell Quality of Life Measurement (ASCQ-Me) Version 2.0 Social Functioning - Short Form questionnaire has a total score ranging from 5-25 with the higher score indicating a healthier status.
Time Frame: Up to 16 weeks
Population: as for outcome 1
Measure: Median (Standard Deviation); unit: score on a scale
Arm/Group | Teduglutide Intervention | Standard of Care Intervention
Number analyzed (Participants) | 6 | 6
score on a scale | 20.5 (5.2) | 20 (7.7)

4. Secondary Outcome: Quality of Life as Measured by the ASCQ-Me® v2.0 Sleep Impact - Short Form
Description: Adult Sickle Cell Quality of Life Measurement (ASCQ-Me) Version 2.0 Sleep Impact - Short Form questionnaire has a total score ranging from 5-25 with the higher score indicating a healthier status
Time Frame: Up to 16 weeks
Population: as for outcome 1
Measure: Median (Standard Deviation); unit: score on a scale
Arm/Group | Teduglutide Intervention | Standard of Care Intervention
Number analyzed (Participants) | 6 | 6
score on a scale | 19.5 (1.3) | 19.5 (4.1)

5. Secondary Outcome: Quality of Life as Measured by the PROMIS Scale v1.2 - Global Health
Description: Patient Reported Outcome Measures Information Systems Global Health has a total score ranging from 10-50 with the higher score indicating a healthier status
Time Frame: Up to 16 weeks
Population: This is a cross-over study. Each participant received both teduglutide intervention and the standard of care intervention for 8 weeks each. 1 participant in the teduglutide arm did not complete the global health questionnaire.
Measure: Median (Standard Deviation); unit: score on a scale
Arm/Group | Teduglutide Intervention | Standard of Care Intervention
Number analyzed (Participants) | 5 | 6
score on a scale | 30 (6.3) | 35 (10.2)

6. Secondary Outcome: Quality of Life as Measured by the PROMIS Scale v1.0 - Gastrointestinal Belly Pain 5a
Description: Patient Reported Outcome Measures Information Systems (PROMIS-GI) Gastrointestinal Belly Pain 5a questionnaire has a total score ranging from 1-25 with the lower score indicating a healthier status
Time Frame: Up to 16 weeks
Population: as for outcome 1
Measure: Median (Standard Deviation); unit: score on a scale
Arm/Group | Teduglutide Intervention | Standard of Care Intervention
Number analyzed (Participants) | 6 | 6
score on a scale | 6.0 (8.2) | 7.5 (6.9)

7. Secondary Outcome: Quality of Life as Measured by the PROMIS Scale v1.0 - Gastrointestinal Diarrhea 6a
Description: Patient Reported Outcome Measures Information Systems (PROMIS-GI) Gastrointestinal Diarrhea 6a questionnaire has a total score ranging from 1-30 with the lower score indicating a healthier status
Time Frame: Up to 16 weeks
Population: as for outcome 1
Measure: Median (Standard Deviation); unit: score on a scale
Arm/Group | Teduglutide Intervention | Standard of Care Intervention
Number analyzed (Participants) | 6 | 6
score on a scale | 8.0 (4.4) | 6.0 (4.0)

8. Secondary Outcome: Quality of Life as Measured by the PROMIS Scale v1.0 - Gastrointestinal Nausea and Vomiting 4a
Description: Patient Reported Outcome Measures Information Systems (PROMIS-GI) Gastrointestinal Nausea and Vomiting 4a questionnaire has a total score ranging from 1-20 with the lower score indicating a healthier status
Time Frame: Up to 16 weeks
Population: as for outcome 1
Measure: Median (Standard Deviation); unit: score on a scale
Arm/Group | Teduglutide Intervention | Standard of Care Intervention
Number analyzed (Participants) | 6 | 6
score on a scale | 3.0 (2.8) | 3.5 (3.3)

9. Secondary Outcome: Quality of Life as Measured by the PROMIS Scale v2.0 - Ability to Participate in Social Roles and Activities - Short Form 8a
Description: Patient Reported Outcome Measures Information Systems (PROMIS) Ability to Participate in Social Roles and Activities - Short Form 8a questionnaire has a total score ranging from 8-40 with the lower score indicating a healthier status
Time Frame: Up to 16 weeks
Population: as for outcome 1
Measure: Median (Standard Deviation); unit: score on a scale
Arm/Group | Teduglutide Intervention | Standard of Care Intervention
Number analyzed (Participants) | 6 | 6
score on a scale | 32.0 (7.8) | 34.0 (13.0)

ADVERSE EVENTS:
Time Frame: Up to 19 months
Groups:
- On Teduglutide: The study is a crossover design. All participants received 8 weeks of daily Teduglutide.
  Teduglutide: Daily 0.05 mg/kg Teduglutide administered subcutaneously.
- On Standard of Care: The study is a crossover design. All participants received 8 weeks of daily Standard of Care Therapy.
  Standard of Care: The standard of care treatment of ECF which includes meticulous wound care, optimizations of nutrition, use of acid-suppression medications and anti-motility agents as per treating physician discretion.
Arm/Group | On Teduglutide | On Standard of Care
All-Cause Mortality (participants affected / at risk) | 0/6 | 0/6
Serious Adverse Events (participants affected / at risk) | 0/6 | 0/6
Other Adverse Events (participants affected / at risk) | 6/6 | 2/6
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | On Teduglutide (N=6) | On Standard of Care (N=6)
Nausea (Gastrointestinal disorders) | 0 (0) | 1 (1)
Vomiting (Gastrointestinal disorders) | 0 (0) | 1 (1)
Stoma hypertrophy (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Pain at fistula site (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Leg Cramps (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Lip Swelling (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Headache (General disorders) | 1 (1) | 0 (0)
Upper Respiratory Infection (Infections and infestations) | 0 (0) | 1 (1)
Right Sided Chest Pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Small Bleeding from Fistula (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
IV Infiltration (Surgical and medical procedures) | 1 (1) | 0 (0)
Increased Creatinine (Renal and urinary disorders) | 1 (1) | 0 (0)
Edema around ostomy site (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Cellulitis (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-06-16): https://cdn.clinicaltrials.gov/large-docs/93/NCT02889393/Prot_SAP_000.pdf